CLINICAL TRIAL: NCT06673810
Title: Effects Of Ankle Weighted Cuffs Training on Kinesthetic Awareness and Toe Walking in Children With Autism Spectrum Disorder.
Brief Title: Effects of Ankle Weighted Cuffs Training in Autism Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/24/0705
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Kinesthetic awareness; Toe walking; Ankle weighted training; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Ankle Weighted Cuffs Training Along with Routine Physical Therapy Exercises
  Interventions: Other: Ankle Weighted Cuffs Training Along with Routine Physical Therapy Exercises
- Control Group (Other): Routine Physical Therapy Exercises
  Interventions: Other: Routine Physical Therapy Exercises

INTERVENTIONS:
Other: Ankle Weighted Cuffs Training Along with Routine Physical Therapy Exercises — Group A will have free ankle weighted cuffs while performing routine physical therapy. These weighted cuffs will be above of the child's ankle and child will be encouraged to perform his/her routine physical activities. Ankle weights will correspond to 2% to 3% of the individual's body weight (sandbags) will be attached at 5 cm above the left and right ankle joints
  Arms: Group A
Other: Routine Physical Therapy Exercises — Group B will perform all the routine physical exercises which include jogging, walk/run interval training, treadmill training and cycling . Intervention period will be of 6 weeks comprising of 3 sessions per week of 30 to 45 minutes per session
  Arms: Control Group

SUMMARY:
Autism spectrum disorders (ASD) are a diverse group of conditions. They are characterized by some degree of difficulty with social interaction, communication and behaviors. Kinesthetic awareness can be defined as how we sense our body and the way it moves. This person might have difficulty understanding where their body is in relation to other objects, thus appearing clumsy, knocking things over, dropping items or misjudging personal space and thus standing too close to others.

DETAILED DESCRIPTION:
The current study will be randomized control trial and data will be collected from (PSRD) pakistan society rehablitation of the disabled. The study will include 44 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will be a parent-confirmed ASD diagnosis from a psychiatrist or licensed psychologist, both male and female children, age between 4 to 14 years. Children with a history of lower limb surgery, a recent (<1 year) ankle sprain and severe behavioral disturbances will be excluded from the study. Experimental group will have ankle weighted cuffs while performing routine physical therapy exercises. Control group will perform routine physical therapy exercises. Outcomes will be analyzed by Limb Position Sense Test and 50 ft walk test. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 25.00.

ELIGIBILITY:
Inclusion Criteria:

* A pre-diagnosed autism spectrum disorder from a psychiatrist or licensed psychologist.
* Both male and female children.
* Age between 4 to 14 years.

Exclusion Criteria:

* Children with a history of lower limb surgery.
* Children with a recent (<1 year) ankle sprain.
* Children presented severe behavioral disturbances, such as aggressive behaviors, self- injurious behaviors, severe motor hyperactivity

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Limb Position Sense Test | 6 weeks
  For the limb-matching test, Participant instructed to keep his eyes closed while the therapist positioned one extremity, and he then was instructed to copy the position with his opposite extremity. Then participant will be asked to replicate 4 positions with his lower extremities while positioned supine on a mat. The limb-matching test positions are described.
  Limb Matching Test Positions
  1. Hip abduction with full knee extension
  2. Hip adduction in neutral
  3. Hip flexion with knee flexion with foot on the mat
  4. Hip and knee flexion at 90° Dynamic Position Sense Movements for Limb Movement Sense Test
  1.Hip circles counterclockwise 2.Hip circles clockwise 3.Active hip abduction and adduction with knee fully extended Intra-class correlations (ICC), which are most often used to express test-retest reliability, were moderate at best, ranging from 0·40 to 0·61 for the four types of position sense tests
50 ft Walk Test | 6 weeks
  The aim of the 50-FWT is to determine the percentage of toe walking performed by each child over a 50ft distance. During the 50-FWT, the children are barefoot to ensure the physical therapist's view of their feet is not obstructed by shoes. To prevent the child from walking past the 50-ft distance, a parent or therapist stands at the end of the walk test to assist in stopping. This allows the physical therapist to read the pedometer value before the child began to move again. The child stands at the start line and the accelerometer is set to 0. Each child ambulates 50 ft. The physical therapist walks at least 6 ft behind the child to assess toe walking while not interfering with gait. The pedometer counts the total number of steps taken during the 50-FWT. The therapist counts the number of steps with initial contact on the toe. The number of toe-walking steps counted by the therapist is divided by the total number of steps counted by the pedometer to get a percentage of toe walking

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Rashida Maqbool, MS*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Society for the Rehabilitation of Disabled, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leyden J, Fung L, Frick S. Autism and toe-walking: are they related? Trends and treatment patterns between 2005 and 2016. J Child Orthop. 2019 Aug 1;13(4):340-345. doi: 10.1302/1863-2548.13.180160. PMID 31489038
- [Background] Armitano-Lago C, Bennett HJ, Haegele JA. Lower Limb Proprioception and Strength Differences Between Adolescents With Autism Spectrum Disorder and Neurotypical Controls. Percept Mot Skills. 2021 Oct;128(5):2132-2147. doi: 10.1177/00315125211036418. Epub 2021 Aug 2. PMID 34340633
- [Background] Guinchat V, Vlamynck E, Diaz L, Chambon C, Pouzenc J, Cravero C, Baeza-Velasco C, Hamonet C, Xavier J, Cohen D. Compressive Garments in Individuals with Autism and Severe Proprioceptive Dysfunction: A Retrospective Exploratory Case Series. Children (Basel). 2020 Jul 13;7(7):77. doi: 10.3390/children7070077. PMID 32668622
- [Background] Valagussa G, Purpura G, Balatti V, Trentin L, Signori A, Grossi E. Quantitative assessment of tip-toe behavior in individuals with autism spectrum disorder and intellectual disability: A cross-sectional study. Autism Res. 2024 Feb;17(2):311-323. doi: 10.1002/aur.3072. Epub 2023 Dec 18. PMID 38108559
- [Background] Washabaugh EP, Augenstein TE, Krishnan C. Functional resistance training during walking: Mode of application differentially affects gait biomechanics and muscle activation patterns. Gait Posture. 2020 Jan;75:129-136. doi: 10.1016/j.gaitpost.2019.10.024. Epub 2019 Oct 21. PMID 31678694